CLINICAL TRIAL: NCT06005766
Title: Does Group-Based Metacognitive Skills Training Reduce Jumping to Conclusions Bias of Patients With Psychotic Disorders in the Context of Forensic Psychiatric Care
Brief Title: The Efficacy of Metacognitive Skills Training in the Context of Forensic Psychiatric Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: Vanha Vaasa Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VVSJYUMCT01
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychotic Disorders; Delusional Disorder; Psychotic Depression
Keywords: Social Cognition; Metacognitive Skills Training; Forensic Psychology; Forensic Psychiatry; Violence
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: There are three groups in the study. One is the intervention group (n=20-25), one consists of patient controls (n=30), and the last one consists of non-patient controls (n=30).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): Patients with a psychosis spectrum disorder participating in the group-based metacognitive skills training and receiving treatment as usual
  Interventions: Behavioral: Metacognitive Skills Training (MCT); Other: Treatment as usual
- Patient controls (Active Comparator): Patients with a psychosis spectrum disorder receiving standard long-term care in the hospital
  Interventions: Other: Treatment as usual
- Non-patient controls (No Intervention): Control group consisting of test subjects without a diagnosis of psychosis spectrum disorder

INTERVENTIONS:
Behavioral: Metacognitive Skills Training (MCT) — The goal of the metacognitive skills training group developed by Moritz and co. is to strengthen the social and metacognitive skills of the patients participating in the group. The group consists of 10 sessions during which exercises and discussion are emphasized. The themes of the group sessions are, for example, jumping to conclusions -bias, empathy, and memory. Detailed information is available from the MCT website (https://clinical-neuropsychology.de/metacognitive_training-psychosis/). Overall there is meta-analysis-level evidence for the moderate effectiveness of MCT on positive symptoms of psychotic illnesses, such as delusions. Prior studies have argued that the unique factor underpinning MCT's efficacy is its impact on various cognitive biases, and that participating in the group especially reduces patients' tendency to jump to conclusions, which is a cognitive style associated with delusions and deficits in social perception and reasoning.
  Arms: Intervention group
Other: Treatment as usual — Medicinal treatment deemed appropriate by the attending physician, psychiatric ward treatment, and others forms of treatment recommended to the patients based on their treatment plans (e.g., work therapy, dialectical behavior therapy, talk therapy)
  Arms: Intervention group; Patient controls

SUMMARY:
Deficiencies in social cognition are part of the core symptomatology of psychotic disorders. And deficiencies in social cognition, the closely related concept of metacognition, and, for example, paranoid attitudes are all associated with violence. The link between social cognition and violence is also observed through rehabilitation, as both group-based Social Cognition Interaction Training (SCIT) and group-based Metacognitive Skills Training (MCT) have reduced violent behavior in patients with psychotic disorders. Thus, a better knowledge of social cognition and its rehabilitation in psychotic disorders can help to reduce risky behavior and to rehabilitate the significant social difficulties often found in psychotic disorders. This research study aims to examine factors underlying the efficacy of group-based MCT.

The goal of the metacognitive skills training group developed by Moritz and partners is to strengthen the social and metacognitive skills of the patients participating in the group. The group consists of 10 sessions during which exercises and discussion are emphasized. The themes of the group sessions are, for example, jumping to conclusions -bias, empathy, and memory. Detailed information is available from the MCT website (https://clinical-neuropsychology.de/metacognitive_training-psychosis/). Overall there is meta-analysis-level evidence for the moderate effectiveness of MCT on positive symptoms of psychotic illnesses, such as delusions. Prior studies have argued that the unique factor underpinning MCT's efficacy is its impact on various cognitive biases, and that participating in the group especially reduces patients' tendency to jump to conclusions, which is a cognitive style associated with delusions and deficits in social perception and reasoning. As delusionality is related to the risk of violence, these results form a logical link between jumping to conclusions, delusionality, and violence.

But the results regarding the effectiveness of MCT are still somewhat conflicting, and studies seem to be of varying quality. Additional longitudinal research and research related to the jumping to conclusion bias are also needed. The hypothesis regarding this study is that the MCT group reduces patients' tendency to jump to conclusions. These reductions are presumed to be associated in one-year follow-up with fewer mood symptoms, delusions, paranoia, and more psychological flexibility.

DETAILED DESCRIPTION:
Based on their multi-professional treatment plan in the Vanha Vaasa hospital, participation in the MCT group intervention is offered to patients who could benefit from it. The intervention under investigation is part of the standard care of the hospital. Participation does not prevent participation in other forms of rehabilitation, and patients can participate in the group even if they don't participate in the study. Being part of the control group does not prevent participation in the intervention group, but being part of the control group might delay participation. When these are in conflict, treatment takes precedence over research.

Data is collected until the sample size is satisfactory (at least 20 to 25 patients). Patients in the MCT condition are compared to patients (n=30) and controls (n=30) measured with a psychological test battery not completing the group. The test battery is the same for all the groups. It consists of valid tasks measuring neurocognition, social cognition, and psychiatric symptoms and a task for measuring the tendency to jump to conclusions. Patients in the group condition are tested before the group and nine months after the group has concluded. For both control groups testing interval is one year.

The comparison between the groups (intervention group, patient controls, and non-patient controls) is done by comparing the rate of change in the tendency to jump to conclusions. This comparison is done with regression analysis. If minor differences and equal variances are assumed (delta of slope 0.1), the power of the comparison is around 0.57. If larger differences are assumed (delta of slope 0.5), the power of the comparison approaches 1. In a previous study, a medium-sized comparative difference between patients in MCT condition and patients in cognitive remediation condition was found.

To avoid problems with multiple testing, the differences in magnitudes of mood symptoms, delusions, paranoia, and psychological flexibility after the delay are assessed with MANOVA. In a recent meta-analysis, the observed effect of MCT on delusions was high medium (g=0.69). The observed effect on negative symptoms was small but significant (g=0.23). Consequently, the expected power of the MANOVA ranges from 0.48 to 0.99. Direct comparisons are made with discriminant analysis with identical power estimates. Univariate ANOVAs can also be used, but with much worse power estimates, when controlling for multiple testing.

ELIGIBILITY:
Inclusion Criteria (patients):

* Willingness to participate in a scientific study
* Diagnosis of a psychosis spectrum disorder
* Finnish language skills due to questionnaires and psychological tests being in Finnish

Exclusion Criteria (patients):

* Psychosis that severely deteriorates the ability to function
* Cognitive problems that severely deteriorate the ability to function
* Guardianship established for personal matters

Inclusion Criteria (non-patient controls):

* Willingness to participate in a scientific study
* Self-assessed sufficient Finnish language skills due to questionnaires and psychological tests being in Finnish

Exclusion Criteria (non-patient controls):

* Diagnosis of a psychosis spectrum disorder
* Cognitive problems that severely interferes with functioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Jumping to conclusions bias | For the intervention group, the measurement is done before the group and nine months after completion. For the control groups, the time interval is one year.
  The bias is measured using a revised version of the beads task. This is a test of optimal performance, meaning that both low and high scores can be problematic.

SECONDARY OUTCOMES:
Paranoia and psychotic experiences | For the intervention group, the measurement is done before the group and nine months after completion. For the control groups, the time interval is one year.
  Paranoia and psychotic experiences assessed with the Symptoms Checklist 90 self-report questionnaire. The scale for paranoia goes from 0 to 24 with higher scores meaning worse outcome. The scale for psychotic experiences goes from 0 to 40 with higher scores meaning worse outcome
Mood symptoms | For the intervention group, the measurement is done before the group and nine months after completion. For the control groups, the time interval is one year.
  Mood symptoms assessed with Symptoms Checklist 90 self-report questionnaire. The sum for scales measuring depression and anxiety goes from 0 to 92 with higher scores meaning worse outcome.
Psychological flexibility | For the intervention group, the measurement is done before the group and nine months after completion. For the control groups, the time interval is one year.
  Psychological flexibility assessed with the the comprehensive assessment of acceptance and commitment therapy processes - Short Form (CompACT-8) self-report questionnaire. The total CompACT score ranges from 0-48, with higher scores indicating greater psychological flexibility: The ability to attend and adapt to situational demands in the pursuit of personally-meaningful longer-term goals.

CONTACTS AND LOCATIONS:
Overall Officials: Raimo Lappalainen, PhD, Principal Investigator — University of Jyvaskyla
Locations (1):
- Vanha Vaasa Hospital, Vaasa, Finland

IPD SHARING:
Plan to Share IPD: Yes
Ownership of the data will reside with the University of Jyväskylä and Vanha Vaasa Hospital. The data are managed by the Ph.D. student, the PI, and the rest of the research team. Other researchers can use the data; however, it requires a research plan and the permission of the research team. Principally, the Ph.D. student, the PI, or someone from the research team will be one of the co-authors in all publications written from the data.